CLINICAL TRIAL: NCT01628796
Title: Ultrasound Measurement of the Acromio-clavicular Joint and Injection of Standard Contrast Material Into the Joint Under Ultrasonic Control
Brief Title: Ultrasound Examination and Guided Injection Into the Acromio-clavicular Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, gordon edelson, Professor of Orthopedic Surgery, The Baruch Padeh Medical Center, Poriya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-2012.CTIL
Record Dates: First submitted 2012-06-19; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis of Acromioclavicular Joint
MeSH Terms: interventions — Contrast Media; iomeprol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: contrast material injection — using ultrasound to locate ac joint and injecting contrast material to ensure that the dye is actually in the joint
  Other Names: iomeron 350

SUMMARY:
Is it possible to improve the accuracy of injection into the acromio-clavicular joint with the use of ultrasound?

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years with AC joint degenerative changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
ultrasound controlled injection of contrast material into the AC joint followed by standard x-ray | outcome assessed at the time of the injection (1 day)
  standard x-ray will be taken after the contrast dye has been injected into the joint to see whether it has successfully been placed into the joint.